CLINICAL TRIAL: NCT04228497
Title: Ultrasound Assessment of Gastric Residual Volume in Children Scheduled for Elective Surgery After Clear Fluids Fasting for One Versus Two Hours; a Comparative Study
Brief Title: Ultrasound Assessment of Gastric Residual Volume in Children Scheduled for Elective Surgery After Clear Fluids Fasting for One Versus Two Hours: a Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MD-87-2019
Record Dates: First submitted 2020-01-11; First posted 2020-01-14 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Gastric Emptying
Keywords: Gastric residual volume; children; ultrasound; fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clear fluids fasting for one hour (Active Comparator): children fasting for 6 to 8 hours will be allowed to drink 3 mL/kg of apple juice to a maximum of 250 ml one hour before surgery
  Interventions: Device: gastric ultrasound; Other: the clear fluid intake
- clear fluids fasting for two hours (Placebo Comparator): children fasting for 6 to 8 hours will be allowed to drink 3 mL/kg of apple juice to a maximum of 250 ml two hours before surgery
  Interventions: Device: gastric ultrasound; Other: the clear fluid intake

INTERVENTIONS:
Device: gastric ultrasound — Children in both groups will be scanned in two positions: supine position and right lateral position (RLP) one and two hours following the clear fluid intake and before admission to the operation room in groups 1 and 2 respectively. Gastric antrum will be located in the sagittal plane with simultaneous identification of left lobe of the liver and the descending abdominal aorta or inferior vena cava.
Other: the clear fluid intake — the clear fluid intake

SUMMARY:
Ultrasound guided comparison of gastric residual volume after clear fluid fasting for one versus two hours in pediatrics scheduled for elective surgery.

DETAILED DESCRIPTION:
Introduction:

The traditional 2-hour clear fluid fasting time was recommended by almost all anesthesia societies [1-3] to decrease the risk of pulmonary aspiration. However, these recommendations are based on historical adult literature [4,5] that may not be applicable to the pediatric population. Moreover, recent studies have shown that these recommendations may not be properly applied, and many children could have been starving for long intervals before surgery with the current guidelines [6-8] which was associated with increased risk of post induction hypotension during surgical preparation [9,10] There is a growing evidence that more liberal clear fluids intake does not result in significant increase in the risk of pulmonary aspiration [11,12] while children may have less thirst, hunger, anxiety, postoperative nausea and vomiting[13-15] also, limiting the fasting time may improve the perioperative inflammatory response in children [16].

Hence, a consensus statement was issued by the Association of Pediatric Anesthetists of Great Britain and Ireland (APAGBI), the European Society of Pediatric Anesthetists and the French-Language Society of Pediatric Anesthesiologists; encouraging clear fluids to be given up to 1 hour before elective general anesthesia [17] which was followed by the Canadian Pediatric Anesthesia Society (CAPS) statement in 2019 [18], however, these statements have not been translated into guidelines to date until further evidence is released.

Gastric residual volume GRV can be used as a preoperative tool for assessment of the risk of perioperative pulmonary aspiration in clinical practice [19]. Many methods have been used to assess gastric volume in pediatrics including nasogastric aspiration [20] , magnetic resonance imaging (MRI) and ultrasound[19,21]. Of these, only ultrasound is of clinical utility because it is simple, bedside, reliable [22], safe tool and allows both qualitative and quantitative assessment of gastric contents [19,23,24].

So, we aim to assess GRV in pediatrics having clear fluids fasting for one hour before elective surgery. We hypothesize that clear fluids fasting for one hour will not result in a clinically significant increase in GRV compared to two hours fasting for children scheduled for elective surgery under general anesthesia.

Methods:

Following approval from Research and Ethics Committee of anesthesia department, Faculty of Medicine, Cairo University. An informed consent will be obtained from parent/care giver prior to commencement of the study.

Inclusion criteria are children aged 3-10 years of both sexes, ASA physical state I and II, scheduled for non-gastrointestinal (GIT) elective day-case surgery under general anesthesia and fasting for 6 to 8 hours or more for solids. Exclusion criteria are parent or care giver refusal, children with gastro-esophageal reflux disease or any disease that impairs gastric motility and children scheduled for emergency surgery.

Patients will be randomly allocated by a computer-generated table into one of the two study groups; the randomization sequence will be concealed in sealed envelopes. Patients and anesthetist doing the ultrasound examination will be blinded to group assignment. The sealed envelopes will be opened in the preparation room by an anesthesia nurse responsible for preparation and offering the fluid to the children depending on the group allocation but not involved in the study data collection. Children fasting for 6 to 8 hours or more for solids only are allowed to drink 3 mL/kg to a maximum of 250 ml of apple juice one hour before surgery in (1-hour group) and two hours before surgery in (2-hours group) .Volume of given "apple juice" will be calculated by a 50 mL scaled clean syringe then poured into a clean cups and offered to the children. Parent/ care giver will be allowed to accompany her/his child during the examination period to alleviate anxiety and ensure compliance of children.

After appropriate time passed, children will be allowed to assess their level of thirst on a 10 cm VAS scale where 0 point is no thirst which will be clarified by laughing face and 10 point is the worst thirst and will be clarified by a crying face. In addition, the parents will grade their child's thirst on a scale of 0-10. Eligible children weight and height will be then measured prior to the examination by a scale and a measuring tape.

Ultrasound examination will be performed using a high frequency (5-10 MHz) ultrasound probe (S-NerveTM; SonoSite Inc., Bothell, WA, USA) or a curvilinear (2-5 MHz) probe as appropriate depending on the child weight and age. Children in both groups will be scanned in two positions: supine position and right lateral position (RLP) exactly one and two hours following the clear fluid intake and before admission to the operation room in groups 1H and 2H respectively. All gastric ultrasound assessments will be completed by the same investigator, who is an anesthetist with 3 years' experience in ultrasound for vascular access and regional anesthesia in pediatric patients. Gastric antrum will be located in the sagittal plane with simultaneous identification of left lobe of the liver and the descending abdominal aorta or inferior vena cava.

According to its shape and contents, the antrum will be considered to be either empty (if it was flat with juxtaposed anterior and posterior walls), fluid-containing (if it was distended, with thin walls and hypoechoic content), or solid-containing (if it was distended with a content of mixed echogenicity).

The antral cross-sectional area (CSA) will be calculated after measuring the two dimensions of the antrum (D1 and D2) according to the following equation: π [D1 × D2] /4, where D1 and D2 are the anteroposterior and craniocaudal diameters, respectively. Measurements will always done from the outer layer of the gastric wall, and all images were obtained between peristaltic contractions. Three measurements will be collected, and average values were used.

The gastric residual volume (GRV) will be calculated using a mathematical model previously validated in the pediatric population [25] as follows :

Gastric residual volume (ml/kg) = [-7.8 + (0.035 ×RLP CSA (mm2) + 0.127 × age (months)]/ body weight (kg)

For quantitative assessment of the risk of aspiration, we will use the classification previously settled by (Van de Putte and Perlas 2014) [24] as follows:

* Low risk of aspiration: children with empty antrum and or children with gastric residual volume less than 1.5 mL/Kg.
* High risk of aspiration: children with solid contents and or children with gastric residual volume more than 1.5 mL/Kg.

If the child has high risk of aspiration, the surgery would be postponed for one hour before another reassessment of the antrum and gastric residual volume.

Anesthetic management:

Upon arrival to the operation room; continuous electrocardiography (ECG), pulse oximetry, non-invasive arterial blood pressure will be applied then general anesthesia will be induced by an experienced pediatric anesthetist who is blinded to the patient group using a controlled rapid sequence induction RSI technique (children in a 20° head up position during preoxygenation and Induction, rapid hypnosis, non-depolarizing muscle relaxant, gentle mask ventilation using Ayres T piece, laryngoscopy, and finally intubation when full motor blockade occurred) [26]. If the patient had no intravenous (IV) cannula; anesthesia will start using titration of 4-8% sevoflurane and 50% air in oxygen using Ayres T piece without positive pressure until the child was put to sleep, peripheral venous cannula will then inserted and anesthesia waill be completed using 0.5-1 mg/kg of propofol. If a patient had an (IV) cannula in place, induction will be performed using 1.5-2.5 mg/kg propofol, in both situations atracurium at a dose of 0.5 mg/kg will be given intravenously to facilitate endotracheal intubation and fentanyl at a dose 2 µg/kg was given to abolish stress response of intubation. The trachea will be then intubated when full motor blockade occurred. Aspiration will be defined as any documentation of vomiting, gastric material in the airway during induction till intubation and confirmation of the endotracheal tube ETT using capnography.

The primary outcome of study will be GRV in right lateral position after one-hour clear fluid intake.

Secondary outcomes are antral cross-sectional area in supine and RLP after one-hour clear fluid intake, antral cross-sectional area in right lateral and supine positions after two hours clear fluid intake, frequency of high risk and low risk of aspiration and qualitative grading for assessment of gastric antrum: three-point as follows: Grade 0: empty antrum, Grade 1: minimal fluid detected in right lateral position only, Grade 2: distended antrum in both semi-sitting and right lateral positions [27]. Incidence of aspiration and or vomiting during induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* • ASA physical state I or II

  * Age 3 to 10 years.
  * Gender: both sexes.
  * Scheduled for non-GIT elective day-case surgery under general anesthesia with endotracheal intubation.

Exclusion Criteria:

* • Parent/ care giver refusal

  * Ages < 3 or > 10 years old
  * Children with gastro-esophageal reflux disease (GORD): either on treatment or under investigation
  * Renal failure, Diabetes mellitus and cerebral palsy patients
  * Esophageal strictures, achalasia or any intestinal disease that may impair the gastric emptying.
  * GIT surgery and neurosurgical patients
  * Emergency surgery

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 226 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
GRV in right lateral position after one-hour clear fluid intake. | one-hour of clear fluid intake

SECONDARY OUTCOMES:
Antral cross-sectional area in right lateral position after one-hour clear fluid intake | one-hour clear fluid intake
Antral cross-sectional area in right lateral and supine positions after two hours clear fluid intake | two hours clear fluid intake
Gastric residual volume in supine position in both groups | one hour after clear fluid intake
Grade of aspiration risk (frequency of high risk and low risk) | one and two hours after clear fluid intake
Qualitative grading for assessment of gastric antrum: three-point grading will be evaluated | one and two hours after clear fluid intake
incidence of aspiration and or vomiting | 10 minutes from induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A Sarhan, MD, Principal Investigator — Lecturer of anesthesia, Cairo university
Locations (1):
- Kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sarhan KA, Hasaneen H, Hasanin A, Mohammed H, Saleh R, Kamel A. Ultrasound Assessment of Gastric Fluid Volume in Children Scheduled for Elective Surgery After Clear Fluid Fasting for 1 Versus 2 Hours: A Randomized Controlled Trial. Anesth Analg. 2023 Apr 1;136(4):711-718. doi: 10.1213/ANE.0000000000006157. Epub 2022 Jul 16. PMID 35881513